CLINICAL TRIAL: NCT01732640
Title: A Phase I/II Study Afatinib/Carboplatin/Paclitaxel Induction Chemotherapy Followed By Standard Chemoradiation In HPV-Negative or High-risk HPV-Positive Locally Advanced Stage III/IVa/IVb HNSCC
Brief Title: A Phase I/II Study Afatinib/Carboplatin/Paclitaxel Induction Chemotherapy In HPV-Negative HNSCC.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual and high levels of toxicity lead to early termination.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Vanderbilt-Ingram Cancer Center (Other); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1266; NA_00074085 (Other: JHMIRB)
Record Dates: First submitted 2012-11-12; First posted 2012-11-26 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Squamous cell carcinoma of the head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Afatinib; Paclitaxel; Carboplatin; Cisplatin; Platinum; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Arm (Experimental): Eligible patients will begin with a 14-day lead-in period with afatinib alone. This will be followed immediately by 2 cycles of induction chemotherapy (IC) with carboplatin AUC 6 IV Day 1, paclitaxel 175mg/m2 IV Day 1, and oral afatinib as a continuous daily dosing. Each cycle is repeated every 21 days. After completion of 2 cycles of IC, patients will be assessed for response by CT/MRI and clinical exam. After the induction, all patients will receive Intensity Modulated Radiation Therapy (IMRT) with weekly cisplatin 40mg/m2 IV. Chemoradiotherapy (CRT) will begin 2-3 weeks after the completion of the second cycle of IC. The patients will be evaluated with a MRI or CT, and FDG PET approximately 12 weeks after completion of CRT.
  Interventions: Drug: Afatinib; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Drug: Afatinib — Afatinib will be supplied as film-coated tablets. Available dosage strengths will be 20, 30, or 40 mg. Tablets will be supplied in HDPE, child-resistant, tamper-evident bottles.
  Other Names: N-[4-[(3-Chloro-4-fluorophenyl)amino]-7-[[(3S)-tetrahydro-3-furanyl]oxy]-6-quinazolinyl]-4(dimethylamino)-2-butenamide
Drug: Paclitaxel — Induction chemotherapy: 175 mg/m2 day 1 every 21 days for 2 cycles (IV infusion as per institutional standard).
  Other Names: TaxolR; NSC 673089
Drug: Carboplatin — Carboplatin is available as a sterile lyophilized powder in single-dose vials containing 50 mg, 150 mg, or 450 mg of carboplatin. Each vial contains equal parts by weight of carboplatin and mannitol. Commercial supplies of carboplatin will be used in this trial.
  Other Names: cis-Diammine(1,1-cyclobutanedicarboxylato)platinum(II)
Drug: Cisplatin — Concurrent chemotherapy: 40 mg/m2 once weekly for 7 cycles (IV infusion as per institutional standard).
  Other Names: Cis-diaminedichloroplatinum Cis-diaminedichloroplatinum (II); diaminedichloroplatinum; cis-platinum; platinum; Platinol; Platinol-AQ; DDP; CDDP; DACP; NSC 119875 R R
Radiation: Intensity Modulated Radiation Therapy — Standard Fractionation 70 Gy /35 fractions at 2 Gy/day for 5 days per week.
  Other Names: IMRT

SUMMARY:
Trial Objectives:

The objective is to investigate the efficacy and safety of afatinib with induction chemotherapy in primary unresected patients with locally advanced, HPV-negative, stage III or IVa/b HNSCC including oral cavity, oropharynx, hypopharynx, or larynx.

Primary Objective Phase I The primary objective of the phase I portion of the trial is to determine the maximum tolerated dose (MTD) or the recommended phase II dose of daily oral afatinib that is safe in combination with carboplatin AUC 6 and paclitaxel 175mg/m2 q 21 days as an induction regimen.

Primary Objective Phase 2 The primary objective of the phase 2 portion of the trial is to estimate the objective tumor response rate and toxicity with induction therapy in patients treated on the afatinib dose determined in Phase I.

Secondary Objectives The secondary objective of phase II is to estimate: 1) the overall response to entire treatment after completion of CRT, 2) progression-free survival (PFS) rate at 2 years, and 3) overall survival (OS) at 2 years.

DETAILED DESCRIPTION:
This is a phase I/phase II prospective multicenter trial to investigate the efficacy and safety of afatinib with induction chemotherapy in primary unresected patients with HPV-negative locally advanced SCC stage III or IVa/b of oral cavity, oropharynx, hypopharynx, or larynx. The primary endpoint is overall response rate after the completion of induction chemotherapy.

Eligible patients will begin with a 14 day lead-in period with afatinib alone. This will be followed immediately by 2 cycles of induction chemotherapy with carboplatin AUC 6 IV, paclitaxel 175mg/m2 day 1, and afatinib as a continuous daily dosing. Each cycle is repeated every 21 days. All patients will receive concurrent chemoradiotherapy beginning 2-3 weeks after the completion of the second cycle of induction chemotherapy (Refer to Study Schema in page 8 of the protocol).

During the period of induction chemotherapy, a complete history and physical (including weight) and tumor assessment by physical examination on Day 1 of each cycle will be performed and documented. Complete blood count with differential and a comprehensive metabolic profile will be performed weekly. After completion of induction chemotherapy, reassessment with blood work, physical exam, CT/MRI of neck and nasopharyngolaryngoscopy will be performed. After the completion of CRT, the patient will have a MRI, CT, or FDG PET approximately 12 weeks after CRT. Follow-up will be standard of care from this point onwards.

Physical exam, blood work and AE assessments will also be frequently performed during entire treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically confirmed diagnosis of squamous cell carcinoma, operable or inoperable tumors, stage III (T3N0-1) and IVA-B (T1-4 N2-3M0 or T4N0-1M0) of oral cavity, oropharynx, hypopharynx and larynx. For patients with oropharynx primary, either HPV negative or HPV positive with a > 10 pack year tobacco history or current smokers are eligible. HPV status should be determined before the enrollment in only non-smokers with oropharynx primary by HPV in-situ hybridization and/or p16 immunostain.
2. Patients must have measurable disease of primary, nodes or both by clinical and radiographic methods per RECIST v1.1..
3. No prior therapy, including surgery with curative intent, chemotherapy, radiation therapy, immunotherapy, EGFR targeted therapies, or any other investigational agents.
4. Age >= 18 years.
5. ECOG performance status 0-1.
6. Patients must have normal hepatic, renal and bone marrow function.

   * Absolute neutrophil count >=1,000/ mm3 Count
   * Platelets >= 100,000/mm3 Count
   * Total serum bilirubin =< 1.5mg/dL Level:
   * AST and ALT =< 2.5 X ULN
   * Alkaline Phosphatase =< 2.5 X ULN
   * Total calculated creatinine clearance >= 60 mL/min
7. Patients with a history of a curatively treated malignancy must be disease-free for at least two years except for carcinoma in situ of cervix and/or non-melanomatous skin cancer.
8. Patients with the following within the last 6 months prior to pre-registration must be evaluated by a cardiologist and/or neurologist prior to entry into the study.

   * Congestive heart failure > NYHA Class II
   * CVA/TIA
   * Unstable angina
   * Myocardial infarction (with or without ST elevation)
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Any prior radiation above the clavicles.
2. Any prior invasive malignancy (unless non-melanomatous resectable skin or the DFS is 2 years or more).
3. History of allergic reactions attributed to compounds of similar chemical or biological composition to afatinib, or other agents used in study.
4. Cardiac left ventricular dysfunction with resting ejection fraction of less than institutional lower limit of normal ( if no lower limit of normal is defined in the institution, the lower limit is 50%)
5. Gastrointestinal tract disease resulting in an inability to take or absorb oral or enteral medication.
6. Baseline significant gastrointestinal symptoms with diarrhoea as a major symptom or a CTCAE Grade >1 diarrhoea of any etiology.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception.
9. Known pre-existing interstitial lung disease (ILD)
10. Pregnant women are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-12; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chung, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Chung CH, Rudek MA, Kang H, Marur S, John P, Tsottles N, Bonerigo S, Veasey A, Kiess A, Quon H, Cmelak A, Murphy BA, Gilbert J. A phase I study afatinib/carboplatin/paclitaxel induction chemotherapy followed by standard chemoradiation in HPV-negative or high-risk HPV-positive locally advanced stage III/IVa/IVb head and neck squamous cell carcinoma. Oral Oncol. 2016 Feb;53:54-9. doi: 10.1016/j.oraloncology.2015.11.020. Epub 2015 Dec 17. PMID 26705063

RESULTS

PARTICIPANT FLOW:
Groups:
- 20 mg Afatinib; 30 mg Afatinib: Eligible patients will begin a 14-day lead-in period with afatinib alone. This will be followed immediately by 2 cycles of induction chemotherapy (IC) with carboplatin AUC 6 IV Day 1, paclitaxel 175mg/m2 IV Day 1, and oral afatinib as a continuous daily dosing. Each cycle is repeated every 21 days. After completion of 2 cycles of IC, patients will be assessed for response by CT/MRI and clinical exam. After the induction, all patients will receive Intensity Modulated Radiation Therapy (IMRT) with weekly cisplatin 40mg/m2 IV. Chemoradiotherapy (CRT) will begin 2-3 weeks after the completion of the second cycle of IC. The patients will be evaluated with a MRI or CT, and FDG PET approximately 12 weeks after completion of CRT.
Period: Overall Study
Arm/Group | 20 mg Afatinib | 30 mg Afatinib
Started | 6 | 3
Completed | 6 | 1
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Eligible patients will begin with a 14-day lead-in period with afatinib alone. This will be followed immediately by 2 cycles of induction chemotherapy (IC) with carboplatin AUC 6 IV Day 1, paclitaxel 175mg/m2 IV Day 1, and oral afatinib as a continuous daily dosing. Each cycle is repeated every 21 days. After completion of 2 cycles of IC, patients will be assessed for response by CT/MRI and clinical exam. After the induction, all patients will receive Intensity Modulated Radiation Therapy (IMRT) with weekly cisplatin 40mg/m2 IV. Chemoradiotherapy (CRT) will begin 2-3 weeks after the completion of the second cycle of IC. The patients will be evaluated with a MRI or CT, and FDG PET approximately 12 weeks after completion of CRT.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
ECOG Status [Count of Participants; unit: Participants] — ECOG of 0 is best value; Normal, no complaints. ECOG of 1 is second best value; Able to carry on normal activities. Minor signs or symptoms of disease.
  Participants
    0 | 6
    1 | 3
Disease Site [Count of Participants; unit: Participants]
  Larynx | 2
  Oropharynx | 6
  Oral Cavity | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Afatinib
Description: The maximally tolerated dose (MTD) was defined as the dose of afatinib in which <2 of 6 patients experience a DLT with the next higher dose having at least 2 of up to 6 patients experiencing a DLT. No dose escalations or de-escalations are permitted within each subject's treatment.
Time Frame: 1 Year (Average)
Measure: Number; unit: mg
Groups:
- All Study Participants: 14-day lead-in period with afatinib alone. This will be followed immediately by 2 cycles of induction chemotherapy (IC) with carboplatin AUC 6 IV Day 1, Eligible patients will begin with a 14-day lead-in period with afatinib alone. This will be followed immediately by 2 cycles of induction chemotherapy (IC) with carboplatin AUC 6 IV Day 1, paclitaxel 175mg/m2 IV Day 1, and oral afatinib as a continuous daily dosing. Each cycle is repeated every 21 days. After completion of 2 cycles of IC, patients will be assessed for response by CT/MRI and clinical exam. After the induction, all patients will receive Intensity Modulated Radiation Therapy (IMRT) with weekly cisplatin 40mg/m2 IV. Chemoradiotherapy (CRT) will begin 2-3 weeks after the completion of the second cycle of IC. The patients will be evaluated with a MRI or CT, and FDG PET approximately 12 weeks after completion of CRT.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
mg | 20

2. Primary Outcome: Objective Tumor Response
Description: Patients were accessed for response by CT/MRI and clinical exam. Partial response was defined as a greater than 30 % reduction in tumor size.
Time Frame: After completion of 2 cycles of induction chemotherapy (at least 8 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- All Study Particpants: Eligible patients will begin with a 4-day lead-in period with afatinib alone. This will be followed immediately by 2 cycles of induction chemotherapy (IC) with carboplatin AUC 6 IV Day 1, paclitaxel 175mg/m2 IV Day 1, and oral afatinib as a continuous daily dosing. Each cycle is repeated every 21 days. After completion of 2 cycles of IC, patients will be assessed for response by CT/MRI and clinical exam. After the induction, all patients will receive Intensity Modulated Radiation Therapy (IMRT) with weekly cisplatin 40mg/m2 IV. Chemoradiotherapy (CRT) will begin 2-3 weeks after the completion of the second cycle of IC. The patients will be evaluated with a MRI or CT, and FDG PET approximately 12 weeks after completion of CRT.
Arm/Group | All Study Particpants
Number analyzed (Participants) | 7
Participants
  Partial Response | 5
  Stable Disease | 2

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Grade 3 or 4 neutropenia (ie. absolute neutrophil count <1000 cells/mm^3) that was associated with a fever>38.5 degrees C or lasting longer than 5 days, grade 3 thrombocytopenia with bleeding or grade 4 thrombocytopenia, and any grade 3 or 4 non-hematologic toxicity per CTCAE criteria which were probably or definitely related to study therapy. During the chemoradiation, an event of stomatitis, pharyngitis, mucositis, or dermatitis was not considered to be a dose limiting toxicity unless it was a grade 4 that did resolve to <grade 2 with a radiation treatment break (not to exceed 10 days) or with withholding chemotherapy (not to exceed 2 weekly doses).
Time Frame: 1 year (average)
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg Afatinib | 30 mg Afatinib
Number analyzed (Participants) | 6 | 3
Participants | 2 | 3

4. Secondary Outcome: Overall Response After Chemoradiation
Description: To estimate the overall response rate after completion of chemoradiation.
Time Frame: 5 Years
Population: Patients were taken off study before the full 5 years could be completed, therefore data was not collected for this outcome measure.
Groups:
- Study Arm: 14-day lead-in period with afatinib alone. This will be followed immediately by 2 cycles of induction chemotherapy (IC) with carboplatin AUC 6 IV Day 1, paclitaxel 175mg/m2 IV Day 1, and oral afatinib as a continuous daily dosing. Each cycle is repeated every 21 days. After completion of 2 cycles of IC, patients will be assessed for response by CT/MRI and clinical exam. After the induction, all patients will receive Intensity Modulated Radiation Therapy (IMRT) with weekly cisplatin 40mg/m2 IV. Chemoradiotherapy (CRT) will begin 2-3 weeks after the completion of the second cycle of IC. The patients will be evaluated with a MRI or CT, and FDG PET approximately 12 weeks after completion of CRT.
  Afatinib: Afatinib will be supplied as film-coated tablets. Available dosage strengths will be 20, 30, or 40 mg. Tablets will be supplied in HDPE, child-resistant, tamper-evident bottles.
  Paclitaxel: Induction chemotherapy: 175 mg/m2 day 1 every 21 days for
Arm/Group | Study Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: 2 Year Progression Free Survival (PFS)
Description: To estimate the 2 year progression free survival.
Time Frame: 2 Years
Population: Patients were taken off study before the full 2 years could be completed, therefore data was not collected for this outcome measure.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Median Overall Survival at 2 Years
Description: To estimate the median overall survival.
Time Frame: 2 Years
Population: as for outcome 5
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Biological Marker Activity of Afatinib
Description: To estimate the biological marker activity of afatinib by serial sampling of tumor and blood samples from patients, and correlate with clinical and pathological response and outcomes. On- and off-target effects of afatinib will be assessed for the biological marker activity.
Time Frame: 5 Years
Population: as for outcome 4
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Activity of Afatinib Based on Serial FLT-PET/CT and DW-MRI
Description: To estimate the activity of afatinib by obtaining serial FLT-PET/CT and DW-MRI, And compare to standard of care CT images (which will be acquired at baseline and at the completion of treatment, and categorized per RECIST criteria) and correlated with response.
Time Frame: 5 Years
Population: as for outcome 4
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Correlate Standard Imaging Pre and Post Treatment
Description: To correlate the response with standard imaging CT/MRI and FDG PET pre and post treatment.
Time Frame: 5 Years
Population: as for outcome 4
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Overall Response After Chemoradiation
Description: To estimate the overall response rate after completion of chemoradiation
Time Frame: 5 years
Population: as for outcome 4
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Only Grade 3-5 Serious Adverse Events were monitored and assessed.
Groups:
- 20 mg Afatinib; 30 mg Afatinib: Eligible patients will begin with a 14-day lead-in period with afatinib alone. This will be followed immediately by 2 cycles of induction chemotherapy (IC) with carboplatin AUC 6 IV Day 1, paclitaxel 175mg/m2 IV Day 1, and oral afatinib as a continuous daily dosing. Each cycle is repeated every 21 days. After completion of 2 cycles of IC, patients will be assessed for response by CT/MRI and clinical exam. After the induction, all patients will receive Intensity Modulated Radiation Therapy (IMRT) with weekly cisplatin 40mg/m2 IV. Chemoradiotherapy (CRT) will begin 2-3 weeks after the completion of the second cycle of IC. The patients will be evaluated with a MRI or CT, and FDG PET approximately 12 weeks after completion of CRT.
Arm/Group | 20 mg Afatinib | 30 mg Afatinib
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg Afatinib (N=6) | 30 mg Afatinib (N=3)
Gr. 4 Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gr. 3 Elevated ALT (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gr. 3 Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Gr. 3 Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gr. 3 Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gr. 3 Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Gr. 3 Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Gr. 4 Sepsis (Infections and infestations) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Slow accrual and high levels of toxicity lead to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No